CLINICAL TRIAL: NCT04480138
Title: A Phase II, Multicenter, Open-label, Randomized, Comparator Controlled Study to Evaluate the Efficacy and Safety of Pegylated Interferon - α2b in the Treatment of Adult Patients Diagnosed With SARS-CoV2 (COVID-19)
Brief Title: Pegylated Interferon - α2b With SARSCoV- 2 (COVID-19)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to non availability of eligible subjects and slow recruitment
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEGI.20.003
Record Dates: First submitted 2020-07-20; First posted 2020-07-21 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2021-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pegylated Interferon-α2b + Standard of care (Experimental): Test :- Pegylated Interferon-α2b + Standard of care (SOC)
  Pegylated Interferon-α2b-Initial 1 mcg/kg will be administered on day 1. After safety evaluation of first dose, next dose (second dose) 1 mcg/kg on day 8 will be administered along with the recommended standard of care at the time of conduct of trial.
  Interventions: Drug: Pegylated Interferon-α2b; Other: Standard of Care
- Standard of Care (Active Comparator): Control: Standard of care
  Standard of care treatment will be provided as per regulatory recommendation and approval.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Pegylated Interferon-α2b — 1 mcg/kg on day 1 and day 8 after safety evaluations.
  Arms: Pegylated Interferon-α2b + Standard of care
Other: Standard of Care — Standard of care as per local authority

SUMMARY:
This is a phase II, multicenter, open-label, randomized, comparator-controlled study to evaluate the efficacy and safety of Pegylated Interferon -α2b in the treatment of adult patients diagnosed with SARS-CoV2 (COVID-19).Initial 1 mcg/kg of Pegylated Interferon-α2b will be administered on day 1. After safety evaluation of first dose, next dose (second dose) 1 mcg/kg on day 8 will be administered with recommended standard care during the trial.

DETAILED DESCRIPTION:
This is a phase II, multicenter, open-label, randomized, comparator-controlled study to evaluate the efficacy and safety of Pegylated Interferon -α2b in the treatment of adult patients diagnosed with SARS-CoV2 (COVID-19).Moderate COVID-19 subjects will be randomly assigned to receive test arm or reference arm in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to comprehend and willingness to sign a written ICF for the study.
2. Male or non-pregnant females, ≥18 years of age at the time of enrolment.
3. Understands and agrees to comply with planned study procedures.
4. Agrees to the collection of pharyngeal swabs and blood sample as per protocol.
5. Has laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay in any specimen within one week
6. Patients with SpO2 > 93% and respiratory rate <30 breaths/min.
7. Illness of any duration, and at least one of the following:

   1. Radiographic infiltrates by imaging (chest x-ray)
   2. Clinical assessment (evidence of rales/crackles or other clinical symptoms on exam).
8. Women of childbearing potential must agree to use at least one primary form of contraception

Exclusion Criteria:

1. ALT/AST >5 times the upper limit of normal.
2. Patients with respiratory rate <20 breaths/min and normal SpO2 with confirmed SARS-CoV-2 infection as determined by PCR (Mild COVID-19 subjects).
3. Patients with respiratory rate ≥30 breaths/min and SpO2 at rest ≤93% (Severe COVID-19 subjects).
4. Stage ≥4 severe chronic kidney disease or requiring dialysis (i.e. eGFR <30 mL/min/1.73 m2).
5. Pregnant or breast feeding.
6. Allergy to any study medication or usage of test drug during last 14 days prior to screening
7. Severe co-morbidity (e.g. uncontrolled hypertension and uncontrolled DM, systemic disease which affect the vital organs severity, immunocompromised patients etc.) as per investigator's assessment.
8. Comorbid condition like myocardial infarction or heart failure within 90 days of recruitment.
9. Prolong QT interval (>450 ms).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Change in Clinical status of subject on a 7-point ordinal scale | Week 2
  1. Not hospitalized, no limitations on activities.
  2. Not hospitalized, limitation on activities.
  3. Hospitalized, not requiring supplemental oxygen.
  4. Hospitalized, requiring supplemental oxygen.
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices.
  6. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
  7. Death.

SECONDARY OUTCOMES:
PCR test | Week 2 and Week 4
  PCR for SARS-CoV-2 in pharyngeal swab
Supplemental Oxygen | Week 2 and Week 4
  Occurrence of supplemental Oxygen
Mechanical Ventilation | Week 2 and Week 4
  Occurrence of Mechanical Ventilation
Incidence of Treatment-Emergent Adverse Events | Week 2 and Week 4
  Occurence of Adverse events
C-reactive protein (CRP) | Week 2 and Week 4
  Inflammatory Biomarker
Interleukin 6 (IL-6) | Week 2 and Week 4
  Inflammatory Biomarker
D-dimer | Week 2 and Week 4
  Inflammatory Biomarker
Interferon gamma | Week 2 and Week 4
  type II class of interferons
Ferritin | Week 2 and Week 4
  proteins
TNF alpha | Week 2 and Week 4
  Inflammatory Biomarker
Interleukin 1-β | Week 2 and Week 4
  Inflammatory Biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Dr Deven Parmar, MD, Study Director — Cadila Healthcare Ltd.
Locations (2):
- Mexico (2):
  - Avant Sante site 2, Zapopan, Jalisco
  - Avant Sante Site 1, Monterrey

IPD SHARING:
Plan to Share IPD: No